CLINICAL TRIAL: NCT01916343
Title: Design of a Comprehensive Evidence-Based Laparoscopy Curriculum for Gynecology Residents
Brief Title: Laparoscopic Gynecology Curriculum for Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12-159
Record Dates: First submitted 2013-06-19; First posted 2013-08-05 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Hysterectomy for Abnormal Uterine Bleeding
Keywords: Laparoscopy; Surgical skills; Team training; Obstetrics and Gynecology; Curriculum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Laparoscopic Curriculum (Experimental): Residents will perform a salpingectomy in the operating room, which will be video-recorded through the laparoscopic camera. The residents in the intervention group will then complete the salpingectomy at the conclusion of the curriculum. Following the completion of the curriculum, residents in the intervention group will undergo a multiple-choice examination as well as a repeat skills examination.
  Interventions: Procedure: Study Laparoscopic Curriculum
- Standard Clinical Education (No Intervention): Residents will perform a salpingectomy in the operating room, which will be video-recorded through the laparoscopic camera. The standard clinical education residents will perform the procedure as per standard of care.

INTERVENTIONS:
Procedure: Study Laparoscopic Curriculum
  Arms: Study Laparoscopic Curriculum

SUMMARY:
Gynecologists are currently using laparoscopy to perform many surgeries traditionally approached by laparotomy. The technical skills required for laparoscopic surgery are different than the skills required for laparotomy, causing a prolonged learning curve. Currently there is no standardized laparoscopy curriculum for gynecology residents. This study aims to develop a specific evidence-based surgical skills gynecologic curriculum that could be instituted in residency programs at a national and international level. The investigators will then validate the curriculum using Obstetrics and Gynecology residents through a cognitive examination, a technical skills examination, and a video recording of performance in the operating room.

HYPOTHESIS: The investigators aim is to design a standardized evidence-based comprehensive laparoscopic curriculum that focuses on cognitive knowledge, surgical skills, and team training exercises. The investigators hypothesize that residents in the experimental curriculum-trained group will perform better than the residents in the traditional residency curriculum-trained group on a cognitive examination, a technical skills examination, and in the operating room. The operating room performance will be judged by blinded experts on a previously validated evaluation tool.

ELIGIBILITY:
Inclusion Criteria:

* Novice residents (defined as having performed less than 10 laparoscopic salpingectomies)
* Patients undergoing uncomplicated right-sided salpingectomies prophylactically at the time of laparoscopic hysterectomy, laparoscopic salpingo-ophorectomies, or laparoscopic-assisted vaginal hysterectomies.

Exclusion Criteria:

* Residents who have performed more than 10 laparoscopic salpingectomies
* Residents in PGY3 or higher
* Patients with multiple prior abdominal surgeries, high BMI, significant adnexal pathology, and extensive endometriosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Technical Performance Score | 9 months
  Technical performance score will be assessed via a previously validated tool known as the OSA-LS (Objective Structured Assessment of Laparoscopic Salpingectomy), with the score received on the OSA-LS being equivalent to their technical score. The OSA-LS is based on the OSATS9, along with a rating scale that has been modified for laparoscopic cholecystectomy. The latter was developed by the primary investigator, Dr. Teodor Grantcharov, and consists of both a reduced global rating scale (GRS) made suitable for laparoscopic surgery, along with a task-specific rating scale known as the operative component rating scale (OCRS). Previously in a pilot study, ten video recorded operations were assessed in order to standardize assessments and to make adjustments to the overall scale. Residents will be video recorded performing a salpingectomy in the operating room. These recordings will be then be scored as per the OSA-LS, by a blinded observer in order to generate an overall assessment.

SECONDARY OUTCOMES:
Cognitive Test Scores | 5 months
  The cognitive training component of the curriculum will consist of of self-directed reading and video-based learning. Participants will learn theoretical principals and management of post operative complications due to laparoscopic gynecologic surgery and watch videos of gynecologic procedures with an expert facilitator.
Surgical Skills | 5 months
  To determine if the proposed laparoscopic curriculum will improve resident scores assessed by cognitive and technical skills examination.

CONTACTS AND LOCATIONS:
Overall Officials: Teodor Grantcharov, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Larsen CR, Grantcharov T, Schouenborg L, Ottosen C, Soerensen JL, Ottesen B. Objective assessment of surgical competence in gynaecological laparoscopy: development and validation of a procedure-specific rating scale. BJOG. 2008 Jun;115(7):908-16. doi: 10.1111/j.1471-0528.2008.01732.x. PMID 18485171